CLINICAL TRIAL: NCT02783339
Title: Evaluation of Safety and Performance of the Neuroform AtlasTM Stent System for Intracranial Aneurysm Treatment - Post Market Clinical Follow-up
Brief Title: Neuroform Atlas Stent for Intracranial Aneurysm Treatment
Acronym: ATLAS EU PMCF
Status: Completed | Type: Observational
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: T4032
Record Dates: First submitted 2016-05-23; First posted 2016-05-26 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Intracranial Aneurysm
Keywords: Next Generation Neuroform Stent System; Intracranial; Stent system; Saccular aneurysm; Stent assisted coiling
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to demonstrate effectiveness and safety of the NeuroForm Atlas stent system for use in patients requiring stent assisted intracranial aneurysm treatment.

DETAILED DESCRIPTION:
The study is a prospective, multicenter, open-label, single arm post market follow-up registry designed to demonstrate the potential treatment of intracranial, saccular aneurysms with the Next Generation Neuroform Stent System. The study will evaluate the permanent morbidity and mortality rate within the 12 to 16 months following the procedure. The study will evaluate as well the percent occlusion of the treated target lesion on angiography in the absence of retreatment, or parent artery stenosis at the target location at 12 to 16 months. Subjects with documented saccular aneurysms arising from a parent artery may potentially benefit from stent assisted coiling, provided they meet the other eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has an intracranial aneurysm for which an endovascular treatment requiring stent assisted intracranial aneurysm coiling has been decided by the site investigator
2. Patient or legal representative is willing and able to provide written informed consent
3. Patient is willing able to comply with scheduled visits and examinations per protocol requirements

Exclusion Criteria:

1. Patient that is younger than 18 years old at the time of entry into the study
2. Patient with mRS > 3
3. Patient has a saccular ruptured aneurysm < 3 months
4. Patient has a fusiform aneurysm
5. Treatment of several aneurysms during the same procedure, except adjacent aneurysms treated with the same stent
6. Planned treatment of other aneurysm in the same vascular territory within the study time period
7. Patient with severe vasospasm that does not respond to pharmacological therapy
8. Aneurysm associated with an arteriovenous malformation, or any other lesion that could lead to hemorrhagic complications
9. Pregnant woman or child feeding
10. Any condition which will not allow the patient to comply with the necessary follow-up for this study (medical condition, patient leaving abroad)
11. Patient with confirmed allergy to nickel titanium (Nitinol)
12. Patient in whom antiplatelet and/or anticoagulation therapy is contraindicate
13. Patient for whom angiography and other examinations show that access to the target cerebral aneurysm by the stent may be impossible because of anatomical features
14. Patient for whom angiography and MRA/MRI is contraindicated
15. Patient with target aneurysm previously treated with a stent -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Registration of patients who are willing to participate in this ATLAS PMCF registry and assuming they meet all of the inclusion/exclusion criteria and provided written informed consent should be recorded prior to implantation of the Neuroform Atlas Stent to ensure data capture on all enrolled and treated patients in this post-market evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
permanent morbidity rate defined as any major ipsilateral stroke or neurolgocial death within 12 to 16 months following the procedure | 16 Months
mortality rate within 12 to 16 months following the procedure | 16 Months

SECONDARY OUTCOMES:
Complete aneurysm occlusion rate of the treated target lesion on 16 month imaging | 16 months
  Measured by the Raymond Scale Class 1,2,3 with imaging at 12 to 16 months
New or worsening major ipsilateral stroke as measured by NIHSS and mRS | 16 months
Subarachnoid hemorrhage rate | 16 months
Aneurysm Rupture rate | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Houdart, MD, PhD, Principal Investigator — Hopital Lariboisière
Locations (11):
- France (6):
  - CHU Pellegrin, Bordeaux
  - CHU Hôpital cavale Blanche, Brest
  - Hôpital Gui de Chauliac, Montpellier
  - CHU Lariboisière, Paris
  - La Fondation Rothschild, Paris
  - CHU Bretonneau, Tours
- Germany (4):
  - Klinikum Augsburg, Augsburg
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Universitätsklinikum Knappschaftskrankenhaus Bochum, Bochum
  - Universität zu Lübeck, Lübeck
- Univerzitná nemocnica Martin, Martin, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lefevre PH, Schramm P, Kemmling A, Barreau X, Marnat G, Piotin M, Berlis A, Wanke I, Bonafe A, Houdart E; ATLAS EU PMCF Investigators. Multi-centric European post-market follow-up study of the Neuroform Atlas Stent System: primary results. J Neurointerv Surg. 2022 Jul;14(7):694-698. doi: 10.1136/neurintsurg-2021-017849. Epub 2021 Sep 2. PMID 34475253